CLINICAL TRIAL: NCT06514820
Title: EXercise Magnetic Resonance Imaging in Patients With Obesity aSsociated Heart failURe With Preserved Ejection Fraction (EXPOSURE) Study
Brief Title: Exercise Magnetic Resonance Imaging in Patients With Obesity Associated Heart Failure
Acronym: EXPOSURE
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: EXPOSURE study
Record Dates: First submitted 2024-07-03; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: Epicardial fat; HFpEF; Exercise MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To aim of the EXPOSURE study is to investigate the effects of epicardial fat on cardiac function, pericardial constraint and pulmonary artery vasodilatation using cardiac magnetic resonance (CMR) imaging at rest and during exercise stress testing in patients with HFpEF.

DETAILED DESCRIPTION:
The EXPOSURE study investigates the effects of epicardial fat on ventricular interdependence at peak exercise. Epicardial fat, the visceral fat situated directly adjacent to the heart, seems involved in the pathophysiology of heart failure with preserved ejection fraction (HFpEF). It has been suggested that an abundance of epicardial fat surrounding the heart within a closed pericardial sac may constrain the heart leading to ventricular interdependence. The study is an investigator initiatied, cross-sectional, observational study, including 50 patients with HFpEF. Patients will be stratified according to high and low epicardial fat volume measured with CMR. The primary outcome parameter is the difference in LV eccentricity index at peak exercise between the two groups. Pre-specified secondary outcome parameters between the subgroups are: 1) VO2-max, 2) LV and right ventricular (RV) diastolic strain rate, 3) slope of early LV/RV filling, 3) left and right atrial reservoir strain and emptying fraction, 4) pulmonary artery distensibility and pulsatility and 5) cardiac output, all at peak exercise. The amount of epicardial fat will be correlated with change in LV eccentricity index from rest to peak exercise, change in LV/RV diastolic strain rate, change in slope of LV/RV filling, change in atrial reservoir strain and emptying fraction, change in pulmonary artery distensibility and pulsatility, and change in cardiac output. All results will be also compared between men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of HF according to the Europeans Society of Cardiology guideline.
2. LV ejection fraction ≥40%.
3. HFA-PEFF score ≥5 or HFA-PEFF score 2-4 in combination with positive stress test (Figure 1).
4. >18 years of age
5. In sinus rhythm
6. Able to perform a bicycle exercise test
7. Willing to sign informed consent

Exclusion Criteria:

1. Body weight >140 kg
2. Atrial fibrillation or other significant arrhythmia during the assessment
3. Contraindications for CMR (e.g. claustrophobia, implanted cardiac devices)
4. Myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft <3 months or untreated severe obstructive coronary artery stenosis
5. More than moderate left-sided valve disease.
6. Complex congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 50 patients with HFpEF, in which the effects of epicardial fat on cardiac function, pericardial constraint and pulmonary artery vasodilatation will be tested using cardiac magnetic resonance (CMR) imaging at rest and during exercise stress testing.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventricular interdependence | Baseline
  the effect of epicardial fat on ventricular interdependence at peak exercise

SECONDARY OUTCOMES:
VO2-max | Baseline
  the effect of epicardial fat on VO2-max at peak exercise
LV/RV diastolic strain rate | Baseline
  the effect of epicardial fat on ventricular diastolic strain rate measured on echocardiography at peak exercise
slope of early LV/RV filling | Baseline
  the effect of epicardial fat on slope of early ventricular filling measured on echocardiography at peak exercise
left and right atrial reservoir strain | Baseline
  the effect of epicardial fat on atrial emptying fraction measured on echocardiography at peak exercise
left and right atrial emptying fraction | Baseline
  the effect of epicardial fat on atrial reservoir strain measured on echocardiography at peak exercise
pulmonary artery distensibility | Baseline
  the effect of epicardial fat on pulmonary artery distensibility measured on echocardiography at peak exercise
pulmonary artery pulsatility | Baseline
  the effect of epicardial fat on pulmonary artery pulsatility measured on echocardiography at peak exercise
cardiac output | Baseline
  the effect of epicardial fat on cardiac output at peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Gorter, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No